CLINICAL TRIAL: NCT03348995
Title: A Prospective Cohort Clinical Trial Evaluating Age as a Risk Factor for Poor Outcomes of Bridge-Enhanced ACL Restoration (BEAR)
Brief Title: The BEAR III Trial for Bridge-Enhanced ACL (Anterior Cruciate Ligament) Restoration
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Miach Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BEAR III Trial
Record Dates: First submitted 2017-11-17; First posted 2017-11-21 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Anterior Cruciate Ligament Injury; Anterior Cruciate Ligament Rupture
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Intervention Model Description: Cohort Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Bridge-Enhanced ACL Restoration (BEAR) (Experimental): The BEAR technique involves surgically placing an absorbable implant (the BEAR Implant) between the torn ends of the ACL, providing a scaffold for the ligament ends to grow into
  Interventions: Device: Bridge-Enhanced ACL Restoration (BEAR)

INTERVENTIONS:
Device: Bridge-Enhanced ACL Restoration (BEAR) — In the BEAR Procedure, surgery is performed to sew the ACL back together and a scaffold is placed between the torn ends at the time of repair.

SUMMARY:
Bridge-Enhanced ACL Restoration (BEAR) is a new procedure being developed to treat patients with ACL injuries. In the BEAR procedure, an implant is placed between the torn ends of the ACL and the patient's own blood is added to the implant to stimulate ligament healing. We propose the current study to determine if older patients do better than younger patients (or vice versa) with this procedure. This is a cohort study designed to determine if age is a risk factor for a worse outcome after a bridge-enhanced ACL repair (BEAR) as defined by an 11.5 point difference on the IKDC Subjective or Objective Knee Evaluation score at two years after surgery. Additional objectives are to determine the effect of age on safety outcomes including infection, graft rejection, and need for further surgical procedures.

DETAILED DESCRIPTION:
The BEAR III study is a cohort study designed to determine if age is a risk factor for a worse outcome after a bridge-enhanced ACL restoration (BEAR) as defined by an 11.5 point difference on the IKDC Subjective or Objective Knee Evaluation score at two years after surgery. Additional objectives are to determine the effect of age on safety outcomes including infection, graft rejection, and need for further surgical procedures.

ELIGIBILITY:
Inclusion Criteria: ACL tear, within 50 days of injury, at least 5% of the ACL attached to the tibia.

-

Exclusion Criteria: Prior surgery on the affected knee, history of knee infection, use of tobacco, use of corticosteroid, chemotherapy, allergy to bovine products or gelatin, history of anaphylaxis, BMI over 35, moderate osteoarthritis.

-

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2018-04-17 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2034-04-17 (Estimated)

PRIMARY OUTCOMES:
International Knee Documentation Committee Subjective Score (IKDC) (Survey) | Time points up to two years
  This is a survey patients complete about how their knee is feeling and functioning. Range is 0 to 100, with 100 indicating no problems and 0 indicating extreme problems.
International Knee Documentation Committee Objective Score (IKDC) (Physical Exam) | Time points up to two years.
  This is an examination performed of the knee. Scores are one of four measures: A (Normal), B (Nearly Normal), C (Abnormal) and D (Severely Abnormal). A is the best outcome and D is the worst.

SECONDARY OUTCOMES:
Knee Injury and Osteoarthritis Score (KOOS) questionnaire | Time points up to two years
  This is a survey with 5 subscales (Pain, Symptoms, Function in Daily Living, Function in Sport and Recreation, and Knee Related Quality of Life). The range of each subscale is 0 to 100, with 100 indicating no problems and 0 indicating extreme problems. The subscales are reported individually and not combined.
Repair Failure | Two years
  The number of times patients develop recurrent knee stability and require another ACL surgery.

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Scripps Health, San Diego, California
  - Florida Orthopedic Institute, Tampa, Florida
  - Emory University School Of Medicine, Atlanta, Georgia
  - Ochsner Sports Medicine Institute, New Orleans, Louisiana
  - MedStar Health Surgery Center of Timonium, Lutherville, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Virtua Health, Marlton, New Jersey
  - Cynthia Chrostek, Providence, Rhode Island
  - Orthopedic Institute of Sioux Falls, Sioux Falls, South Dakota
  - UT Southwestern, Dallas, Texas
  - Inova Sports Medicine, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No